CLINICAL TRIAL: NCT06940024
Title: Comparison of Accuracy of Maxilla Between Virtual Surgical Planning and Conventional Surgical Planning in Bimaxillary Orthognathic Surgery: a Randomized Controlled Trial
Brief Title: Comparison of Accuracy of Maxilla Between Virtual and Conventional Surgical Planning in Bimaxillary Orthognathic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Phuoc Loi, Principal Investigator, Lecturer of Maxillofacial Surgery Department, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 647/HĐĐĐ-ĐHYD
Record Dates: First submitted 2025-03-25; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-06

CONDITIONS: Orthognathic Surgical Procedures; 3D Printing; Splints
Keywords: Orthognathic Surgery; 3D planning; Splints; Accuracy of maxillary postion

STUDY DESIGN:
Intervention Model Description: After determining the desired the maxillary and mandibular position by 3D planning, involved fabricating surgical splints using two different methods:
  * CSP Group (Conventional Resin Occlusal Splint - Control group): Splints were manually fabricated based on P3D movement values. Maxillary landmark points were marked, and the upper jaw cast model was segmented and repositioned to match P3D maxillary to the nearest approximation base on anterior-posterior and superior-inferior changes of these points. The actual movement distances of U1L, U1R, U3L, U3R, U6L, and U6R were recorded as PCM (Planning Cast Model).
  * VSP Group (Virtual Digital Occlusal 3D Print Splint - Interventional group): Digital surgical splints were generated using Dolphin software and a Form 3D printer.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CSP Group (Conventional Resin Occlusal Splint) (No Intervention): Splints were manually fabricated based on 3D planning movement values
- VSP Group (Experimental): Digital surgical splints were generated using Dolphin software and a Form 3D printer
  Interventions: Device: VSP Group

INTERVENTIONS:
Device: VSP Group — Digital surgical splints were generated using Dolphin software and a Form 3D printer
  Arms: VSP Group

SUMMARY:
Study Title Comparison of Maxillary Accuracy Between Virtual and Conventional Surgical Planning in Bimaxillary Orthognathic Surgery: A Randomized Controlled Trial Study Design

* Type: Prospective, single-center, randomized, blinded, case-controlled trial
* Location: National Hospital of Odonto-Stomatology, Ho Chi Minh City
* Period: August 2023 - February 2025
* Sample size: 20 patients
* Ethical approval: Granted by the University of Medicine and Pharmacy at HCMC (Approval No. 647/HĐĐĐ-ĐHYD) Inclusion Criteria
* Patients aged 18-30 years
* Diagnosed with malocclusion requiring bimaxillary orthognathic surgery
* Completed presurgical orthodontic treatment Exclusion Criteria
* Cleft lip/palate, craniofacial syndromes
* Deformities due to trauma, tumors, or iatrogenic causes
* TMJ disorders
* History of previous orthognathic surgery
* Planned multipiece Le Fort I osteotomy Randomization and Blinding
* All patients underwent both 2D and 3D surgical planning.
* Two splints (CSP and VSP) were fabricated for each patient.
* Intraoperative randomization was performed by an OR nurse.
* The surgical team and data analysts were blinded to group allocation.
* Groups were revealed only after data analysis. Groups
* Test group (VSP): 3D virtual planning, simulation, and 3D-printed splints
* Control group (CSP): 2D cephalometric planning, model surgery, conventional resin splints Surgical Procedure
* All patients underwent Le Fort I and BSSO
* Maxilla-first approach with fixation using 4 miniplates
* Mandibular repositioning using final splint and fixed with 2 miniplates per side
* All surgeries performed by a single experienced surgeon Data Collection & Measurements
* CT scans before and 2 weeks after surgery
* Superimposition using Invivo 7.0 software (voxel-based registration)
* Measured landmark changes (A point, ANS, U1, U3, U6) in X (medial-lateral), Y (anterior-posterior), and Z (vertical) directions
* Compared:

  * 2D plan (P2D) vs. 3D plan (P3D)
  * P3D vs. actual postoperative result
  * VSP vs. CSP accuracy Statistical Analysis
* ICC used to test measurement reliability (10 patients, remeasured after 2 weeks)
* Normality tested
* Paired t-test/Wilcoxon for planned vs. actual
* Independent t-test/Mann-Whitney for between-group comparisons
* Significance set at p < 0.05

DETAILED DESCRIPTION:
Materials and Methods Study Design This study was conducted as a prospective, single-center, randomized, and blinded case-controlled trial. The research protocol was reviewed and approved by the Ethics Committee of the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 647/HĐĐĐ-ĐHYD). All participants were fully informed of their treatment options and provided written informed consent prior to enrollment. The study adhered to ethical guidelines for clinical research, ensuring the protection of participants' rights, safety, and confidentiality.

Study Subjects The study was carried out at the National Hospital of Odonto-Stomatology in Ho Chi Minh City between August 2023 and February 2025. Eligible participants were aged 18 to 30 years and diagnosed with malocclusion requiring bimaxillary orthognathic surgery.

Exclusion criteria included:

1. Cleft lip and/or palate or craniofacial syndromes
2. Facial deformities resulting from trauma, tumors, or iatrogenic causes
3. Temporomandibular joint disorders
4. Previous history of orthognathic surgery
5. Indication for multipiece Le Fort I osteotomy A total of 20 patients met the inclusion criteria and agreed to participate. All patients had completed presurgical orthodontic treatment prior to surgery.

Randomization and Blinding Each patient underwent both two-dimensional (2D) lateral cephalometric analysis and three-dimensional (3D) virtual surgical planning preoperatively. For each case, both a conventional surgical splint and a 3D-printed splint were fabricated.

Randomization was performed intraoperatively by an operating room nurse through a simple draw to determine which splint would be used. Allocation was recorded accordingly. The surgical and research teams were blinded to group assignment, with participants identified only as "Group 1" or "Group 2." Group identities (VSP or CSP) were only disclosed after data collection and analysis were complete.

Patients were assigned to two groups:

* Test group (VSP): 3D imaging, virtual osteotomy simulations, and 3D-printed splints
* Control group (CSP): 3D imaging, virtual osteotomy simulations, model surgery, and hand-fabricated resin splints Methods Preoperative Examination and Surgical Planning All patients underwent a full preoperative assessment, including clinical examination, radiographic imaging (panoramic, lateral and posteroanterior cephalograms, and CT scans), 2D cephalometric analysis, intraoral and facial photography, and dental impressions.

Facebow registration and intermaxillary relationship assessment were performed, followed by mounting on a semi-adjustable articulator using the standard Frankfort horizontal plane. Final occlusion was determined by the orthodontist. Dental models were digitized using the Autoscan-DS-EX Pro (Shining 3D) scanner.

Surgical planning was initially based on clinical findings and 2D cephalometric analysis using WebCeph software. Parameters included maxillary dental midline, anteroposterior and vertical positioning of maxillary incisors, and occlusal plane canting determined by the canine and first molar reference points.

3D Simulation

A 3D virtual skull model was constructed using anatomical reference planes for consistent orientation:

* Horizontal plane: through Nasion, parallel to the Frankfort horizontal plane
* Midsagittal plane: through Nasion and Basion, perpendicular to the horizontal plane
* Coronal plane: through Nasion, perpendicular to both horizontal and midsagittal planes The mandible was repositioned into the final occlusion, and the maxillomandibular complex was aligned according to P2D (Planning 2D) parameters derived from 2D analysis. Maxillary landmarks (A point, ANS, U1, U1L, U1R, U3L, U3R, U6L, U6R) were recorded.

Next, refinements were applied using VSP to adjust occlusal plane canting, midline deviation, yaw rotation, and anteroposterior and vertical positioning based on Vietnamese normative standards. These refined landmark positions were recorded as P3D (Planning 3D).

Comparison Between P2D and P3D Differences in landmark movements between P2D and P3D (A point, ANS, U1, U1L, U1R, U3L, U3R, U6L, U6R) were analyzed to assess the discrepancies between 2D and 3D planning methods.

Group Allocation and Splint Fabrication

After determining the final maxillary and mandibular positions, surgical splints were fabricated as follows:

* CSP Group (Conventional Resin Occlusal Splint): Splints were manually fabricated based on P3D values. Landmarks were marked, and the maxillary model was segmented and repositioned to approximate the P3D position based on anterior-posterior and superior-inferior displacements. The actual repositioning distances of U1L, U1R, U3L, U3R, U6L, and U6R were recorded as PCM (Planning Cast Model).
* VSP Group (Virtual 3D-Printed Splint): Surgical splints were digitally generated using Dolphin software and printed using a Formlabs 3D printer.

Surgical Procedures All surgeries were performed by the same experienced maxillofacial surgeon using a standardized maxilla-first approach.

* Maxillary osteotomy was performed first (LeFort I), and the maxilla was positioned using the intermediate splint, with position verified by simulation images. Rigid fixation was performed using four miniplates and screws.
* Mandibular osteotomy followed (BSSO technique), and repositioning was guided by the final splint. Fixation was achieved with two miniplates per side.
* Final verification of skeletal alignment and occlusion was conducted before layered soft tissue closure.
* Intermaxillary fixation was not routinely used, but light elastics were applied as needed.

Postoperative Skeletal Accuracy Analysis Two weeks post-surgery, all patients underwent CT imaging in occlusion with the final splint and before initiation of postoperative orthodontic treatment.

Pre- and postoperative scans were superimposed using voxel-based registration (Invivo 7.0, Anatomage, CA), aligned to non-surgical cranial reference areas using the same reference planes:

* X-axis: medio-lateral (positive = left)
* Y-axis: antero-posterior (positive = forward)
* Z-axis: superior-inferior (positive = downward) Landmark movements (A point, ANS, U1, U1L, U1R, U3L, U3R, U6L, U6R) were recorded as Actual values.

Surgical accuracy was evaluated through:

* Intra-group comparisons: P3D vs. Actual positions for each landmark
* Inter-group comparisons: Discrepancies between VSP and CSP groups Measurement Methods for Accuracy Assessment The intraclass correlation coefficient (ICC) was used to assess measurement reliability. Ten patients were randomly selected and remeasured after two weeks.

Statistical Analysis

* Normality testing was performed for all variables.
* If normally distributed, paired t-tests were used for P3D vs. Actual, and independent t-tests for CSP vs. VSP comparisons.
* If non-normally distributed, Wilcoxon signed-rank and Mann-Whitney U tests were applied.
* A p-value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malocclusion requiring orthognathic surgery

Exclusion Criteria:

* cleft lip and palate congenital abnormalities
* the facial deformities were caused by trauma, tumor, or iatrogenic factors
* temporomandibular joint disorders
* history of previous orthognathic surgery
* patients scheduled for multipiece Le Fort I osteotomy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the anteroposterior, mediolateral, and superoinferior changes of the maxillary landmarks were calculated to assess accuracy and validate the effectiveness of virtual surgical planning | From August 2023 to February 2025
  The accuracy of surgical outcomes was evaluated through: Positional Change of A Point, ANS, maxillary central incisors midpoint (U1), left maxillary central incisor (U1L), right maxillary central incisor (U1R), Maxillary Canines (U3L, U3R), Maxillary First Molars (U6L, U6R) (mm) Comparison of surgical accuracy between Planning and Acutual (mm differences) in each group • Description: The distance differences (in millimeters) between the planned 3D position (P3D) and the actual postoperative position (Actual) of each anatomical landmark was measured using voxel-based registration on superimposed preoperative and postoperative CT scans (2 weeks after surgery) using Invivo 7.0 software.
  Comparison of Surgical Accuracy Between VSP and CSP (mm deviation)
  • Description: The absolute positional deviations (in mm) of each anatomical landmark were compared between the VSP and CSP groups to assess which surgical planning method yielded higher accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- 201A, Nguyen Chi Thanh Street, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen H, Bi R, Hu Z, Chen J, Jiang N, Wu G, Li Y, Luo E, Zhu S. Comparison of three different types of splints and templates for maxilla repositioning in bimaxillary orthognathic surgery: a randomized controlled trial. Int J Oral Maxillofac Surg. 2021 May;50(5):635-642. doi: 10.1016/j.ijom.2020.09.023. Epub 2020 Oct 31. PMID 33131986
- [Background] Schneider D, Kammerer PW, Hennig M, Schon G, Thiem DGE, Bschorer R. Customized virtual surgical planning in bimaxillary orthognathic surgery: a prospective randomized trial. Clin Oral Investig. 2019 Jul;23(7):3115-3122. doi: 10.1007/s00784-018-2732-3. Epub 2018 Nov 15. PMID 30443778
- [Background] Ritto FG, Schmitt ARM, Pimentel T, Canellas JV, Medeiros PJ. Comparison of the accuracy of maxillary position between conventional model surgery and virtual surgical planning. Int J Oral Maxillofac Surg. 2018 Feb;47(2):160-166. doi: 10.1016/j.ijom.2017.08.012. Epub 2017 Sep 23. PMID 28950997
- [Background] Song KG, Baek SH. Comparison of the accuracy of the three-dimensional virtual method and the conventional manual method for model surgery and intermediate wafer fabrication. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Jan;107(1):13-21. doi: 10.1016/j.tripleo.2008.06.002. Epub 2008 Aug 28. PMID 18755612
- [Background] Xu R, Ye N, Zhu S, Shi B, Li J, Lai W. Comparison of the postoperative and follow-up accuracy of articulator model surgery and virtual surgical planning in skeletal class III patients. Br J Oral Maxillofac Surg. 2020 Oct;58(8):933-939. doi: 10.1016/j.bjoms.2020.04.032. Epub 2020 May 20. PMID 32446591